CLINICAL TRIAL: NCT04017026
Title: Survival and Success Rates of 6mm Implants With a Micro-rough Surface After 4.5 - 18.2 Years in Function
Status: Completed | Type: Observational
Sponsor: University of Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 2019_6mm_implants
Record Dates: First submitted 2019-04-03; First posted 2019-07-12 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-09

CONDITIONS: Jaw, Edentulous, Partially; Dental Implant Failed; Implant Complication
Keywords: Short dental implant; Partially edentulous jaw
MeSH Terms: conditions — Jaw, Edentulous, Partially

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- 6 mm implants: Patients were treated with 6mm short implants (Straumann, SLA, SLActive, 4.1 or 4.8 mm in diameter).
  Interventions: Device: Implantation

INTERVENTIONS:
Device: Implantation — Implantation of 6 mm short implants

SUMMARY:
In this retrospective study, approximately 60 patients treated with 6mm short implants (Straumann, SLA (sandblasted, large-grit, acid-etched surface), SLActive (sandblasted, large-grit, acid-etched, hydrophilic surface), 4.1 or 4.8 mm in diameter) will be followed for 4.5-18.2 years. Clinical and radiographic parameters will be assessed in a follow-up examination.

ELIGIBILITY:
Inclusion Criteria:

* Partially or fully edentulous jaw
* Written informed consent

Exclusion Criteria:

* Pregnant women/lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients treated with a 6mm short implant at the University of Bern were recalled for a clinical and radiographic follow-up examination.
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2018-05-09 (Actual); Primary Completion 2019-04-08 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Implant survival rates | 5-18 years
  Survival rates of short dental implants

SECONDARY OUTCOMES:
Radiographic: Annual bone loss | 5-18 years
  Distance from the implant shoulder to the marginal bone.
Clinically: modifying risk factors on implant survival and success | 5-18 years
  Plaque-index
Clinically: modifying risk factors on implant survival and success | 5-18 years
  Sulcus bleeding index
Clinically: modifying risk factors on implant survival and success | 5-18 years
  Probing depth
Clinically: modifying risk factors on implant survival and success | 5-18 years
  Prosthetic reconstruction
Clinically: modifying risk factors on implant survival and success | 5-18 years
  Implant position
Clinically: modifying risk factors on implant survival and success | 5-18 years
  Crown-to-implant ratio
Patient reported outcome measures | 5-18 years
  Visual analog scale (satisfaction between 0 - 100%)
Patient reported outcome measures | 5-18 years
  Oral health impact profile
Implant success rates | 5-18 years
  Success rates of dental implants. Success rates according to Buser et al. 1990.

CONTACTS AND LOCATIONS:
Overall Officials: Vivianne Chappuis, DMD, Study Chair — University of Bern
Locations (1):
- Department for oral surgery of the zmk Bern, University of Bern, Bern, Switzerland